CLINICAL TRIAL: NCT03314948
Title: Ultrasound-Guided Costoclavicular Block in Patients With a BMI > 30
Status: Terminated | Type: Observational
Why Stopped: Due to lack of resources and changes in current practice, the study was terminated
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher B. Robards, Principal Investigator, Mayo Clinic
Other Study IDs: 17-006489
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Researchers are trying to determine if Costoclavicular brachial plexus block (CCBPB) can be successfully performed in patients with a body mass index greater than thirty.

ELIGIBILITY:
Inclusion Criteria:

18 to 80 years old, with American Society of Anesthesiologists physical status I to IV, undergoing elective hand or forearm surgery under a BPB will be enrolled for this study.

Exclusion Criteria:

Patient's refusal, American Society of Anesthesiologist physical status greater than IV, pregnancy, neuromuscular disease, prior surgery on the intraclavicular fossa, nerve injury or neurological disorders, bleeding tendency or evidence of coagulopathy, history of allergy to local anesthetic drugs, skin infection at the site of needle insertion, or contraindication to regional anesthesia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing an elective hand or forearm surgery
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Success rate of costoclavicular brachial plexus block | Within 45 minutes of completion of block placement
  Determine the success rate of the block in patients with body mass index greater than 30. Assess the effectiveness of the block by performing required assessments

SECONDARY OUTCOMES:
Identification of costoclavicular space | during placement of the block
  Describe how the costoclavicular space and its contents are easily identifiable in patients with a body mass index greater than 30. Identify the costoclavicular space by using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Robards, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials